CLINICAL TRIAL: NCT02645786
Title: Cardiac Effects of Thyrotropin Over-Suppression With Levothyroxine in Young Women With Differentiated Thyroid Cancer
Brief Title: Thyrotropin Over-suppression and Heart
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, OHKHYUN RYU, Associate professor, Chuncheon Sacred Heart Hospital
Other Study IDs: 2009-19
Record Dates: First submitted 2015-12-20; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Malignant Neoplasm of Thyroid; Heart Diseases; Thyrotoxicosis on Thyroxine Therapy
Keywords: thyroid neoplasms; heart; thyroxine; thyrotoxicosis
MeSH Terms: conditions — Thyroid Neoplasms; Heart Diseases; Thyrotoxicosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Differentiated thyroid cancer group:
  who received total- or near-total thyroidectomy, and thereafter regularly visited the endocrine out-patient department (OPD) of Chuncheon Sacred Heart Hospital.
  1) age less than 45 years old when receiving total or near-total thyroidectomy, 2) serum level of TSH<0.1 mU/L in the intermediate recurrence-risk or TSH<0.3 mU/L in the low recurrence-risk group13, 14 over 2 years before study entry, 3) receiving TSH suppressive therapy for 5 to 9 years with fixed dose of LT4 more than 2 years before study entry, and 4) no history of structural heart disease, arrhythmia, or cardiac symptoms (palpitation, exertional dyspnea and chest discomfort) during therapy.
- Control: Control group As each DTC patient was enrolled, control subjects were selected from patients who visited endocrinology department for thyroid nodule work-up. The control group had to meet the following criteria
  1) the subject matched to a patient by age (±2 years), sex, and body mass index (BMI) (±2 kg/m2), 2) within the reference range of serum TSH (0.3-4.6 mU/L), 3) no history of structural heart disease, arrhythmia, or cardiac symptoms, 4) no history of comorbid diseases which affect thyroxine metabolism and cardiac structure, including hepatic or renal disease, anemia, and hypertension.

SUMMARY:
The investigators evaluated the cardiac effects of Thyroid-stimulating hormone (TSH) over-suppression in women with differentiated thyroid cancer (DTC) frequently encountered during suppression therapy.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the cardiac effects of TSH over-suppression in women with DTC during TSH suppressive therapy for 5 to 9 years relative to their risk of recurrence.

Methods

1. Patients

   From chart review, the investigators selected 96 female differentiated thyroid cancer patients who received total- or near-total thyroidectomy, and thereafter regularly visited the endocrine out-patient department (OPD) of Chuncheon Sacred Heart Hospital. Majority of papillary thyroid cancer tends to present between 30 and 50 years old and their risk of recurrence is low or intermediate. Menopause also might affect on the cardiovascular risk factors in women. According to guidelines, the dose of thyroxine would be reduced after 10 years of thyroidectomy in DTC patients. Therefore, additional enrollment criteria were as follows: 1) age less than 45 years old when receiving total or near-total thyroidectomy, 2) serum level of TSH<0.1 mU/L in the intermediate -risk or TSH<0.3 mU/L in the low recurrence-risk group, over 2 years before study entry, 3) receiving TSH suppressive therapy for 5 to 9 years with fixed dose of LT4 more than 2 years before study entry, and 4) no history of structural heart disease, arrhythmia, or cardiac symptoms (palpitation, exertional dyspnea and chest discomfort) during therapy. Of the 17 patients who met the criteria, three patients did not consent to this study. Candidates who satisfied all the enrollment criteria took an electrocardiogram to rule out patients with arrhythmia. Finally, 14 DTC patients were enrolled and studied from September 2009 to March 2010. As each patient was enrolled, control subjects were selected from patients who visited endocrinology department for thyroid nodule work-up. The control group had to meet the following criteria: 1) the subject matched to a patient by age (±2 years), sex, and body mass index (BMI) (±2 kg/m2), 2) within the reference range of serum TSH (0.3-4.6 mU/L), 3) no history of structural heart disease, arrhythmia, or cardiac symptoms, 4) no history of comorbid diseases which affect thyroxine metabolism and cardiac structure, including hepatic or renal disease, anemia, and hypertension. All subjects who met the enrollment criteria took an electrocardiogram to rule out arrhythmias. Control subjects were recruited and tested from January 2010 to July 2011. All participants provided written informed consent.
2. Assays

   On the examination day, all participants were prohibited from smoking and consuming caffeine. After a light breakfast and medication, including levo-thyroxine (LT4) in cancer patients, participants visited the hospital before 9 AM. The investigators evaluated the comorbid conditions of the participants. Body weight and height were measured while the participants wore light clothing without shoes. The body mass index (BMI) was calculated as the weight in kilograms divided by the height in meters squared. Their blood pressure was taken after a 10 minute rest period. Subsequently, each subject underwent a 2-dimensional echocardiogram carried out by one examiner. After the cardiac work-up, blood samples were drawn to test of thyroid function. Blood samples were collected in pre-chilled tubes containing EDTA, immediately placed on ice, and promptly centrifuged at 4°C. After separation, plasma was stored at -80°C for the N-terminal pro-brain natriuretic peptide (NT-pro-BNP).

   Serum thyroid function tests were performed by a chemiluminescent immunoassay (UNICELL DXI800, Beckman Coulter, USA). Serum TSH (reference value: 0.3-4.6 mU/L, detection limit: 0.0025 mU/L), free T4 (reference value: 7.0-20.0 pmol/L), and free T3 (reference value: 4.0-5.9 pmol/L) were measured. Plasma NT-pro-BNP measurements were done using chemiluminescent immunoassay method (Roche E170, Roche diagnostics, Germany)
3. Echocardiography

Comprehensive transthoracic echocardiography was performed using commercially available equipment (IE33, Philips Medical System, Andover, Massachusetts). Standard 2-dimensional measurements were obtained as recommended by the American Society of Echocardiography (ASE) in the left lateral position. Left atrial volume index was measured by the biplane area-length method. Left ventricular (LV) mass was calculated using the following equation: LV mass = 0.8 (1.04 { [LVIDd + PWTd + IVSd]3 - [LVIDd]3 } )+ 0.6, where LVID is LV end-diastolic dimension, PWT is posterior wall thickness, IVS is interventricular septal wall thickness, and d is diastole. Tissue Doppler-derived early diastolic mitral annular velocity (e') and late diastolic mitral annular velocity (a') were measured from the septal corner of the mitral annulus in the apical 4-chamber view. To evaluate the global longitudinal strain (GLS) of the left ventricle, echocardiographic images were obtained at the apical 4-chambers view and the strain was analyzed based on routine DICOM (Digital Imaging and Communications in Medicine) data sets using software (2D Cardiac Performance Analysis, TomTec, Munich, Germany). A region of interest was manually placed on the endocardial and epicardial borders. The echocardiographic data were gathered and analyzed by 2 experienced echocardiographers who were unaware of any corresponding clinical data.

Statistical analysis Data were reported as means and standard deviation (SD). For the comparison of means between groups, we used the Mann-Whitney test because the sample size was small (n=14 for each group).

All P values calculated are two-tailed and considered significant at P < 0.05. All statistical analysis was performed using SPSS 20.0 software (SPSS Inc, Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

* thyroid cancer group

  1. age less than 45 years old when receiving total or near-total thyroidectomy,
  2. serum level of TSH<0.1 mU/L in the intermediate -risk or TSH<0.3 mU/L in the low recurrence-risk group over 2 years before study entry,
  3. receiving TSH suppressive therapy for 5 to 9 years with fixed dose of LT4 more than 2 years before study entry, and
  4. no history of structural heart disease, arrhythmia, or cardiac symptoms (palpitation, exertional dyspnea and chest discomfort) during therapy.
* control group

  1. the subject matched to a patient by age (±2 years), sex, and body mass index (BMI) (±2 kg/m2),
  2. within the reference range of serum TSH (0.3-4.6 mU/L),
  3. no history of structural heart disease, arrhythmia, or cardiac symptoms,
  4. no history of comorbid diseases which affect thyroxine metabolism and cardiac structure, including hepatic or renal disease, anemia, and hypertension.

Exclusion Criteria:

* who had arrhythmia in electrography or history of cardiac disease

Ages: 32 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female differentiated thyroid cancer patients who received total- or near-total thyroidectomy, and thereafter regularly visited the endocrine out-patient department (OPD) of Chuncheon Sacred Heart Hospital. Finally, 14 DTC patients were enrolled and studied from September 2009 to March 2010. As each patient was enrolled, control subjects were selected from patients who visited endocrinology department for thyroid nodule work-up. All subjects who met the enrollment criteria took an electrocardiogram to rule out arrhythmias.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2009-09; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
comparison of cardiac fucntion and structure between groups | measure cardiac function and struture at 2009 in case (DTC group) and at 2010 in control group
  In DTC group, the investiagtors measured cardiac function and structure by echocardiography at 2009 (receiving TSH suppressive therapy for 5 to 9 years after thyroidectomy). As each DTC patient was enrolled, control subjects were selected from persons who visited endocrinology department for thyroid nodule work-up. The control group had to meet the following criteria: 1) the subject matched to a patient by age (±2 years), sex, and body mass index (BMI) (±2 kg/m2), 2) within the reference range of serum TSH (0.3-4.6 mU/L), 3) no history of structural heart disease, arrhythmia, or cardiac symptoms, 4) no history of comorbid diseases which affect thyroxine metabolism and cardiac structure, including hepatic or renal disease, anemia, and hypertension.The cardiac function and structure were evaluated by echocardiography at 2010.

SECONDARY OUTCOMES:
comparison of heart rate between groups | measure heart rate at 2009 in case (DTC group) and at 2010 in control group.
  In DTC group, the investiagtors measured heart rate at 2009 (receiving TSH suppressive therapy for 5 to 9 years after thyroidectomy). As each DTC patient was enrolled, control subjects were selected from persons who visited endocrinology department for thyroid nodule work-up. The control group had to meet the following criteria: 1) the subject matched to a patient by age (±2 years), sex, and body mass index (BMI) (±2 kg/m2), 2) within the reference range of serum TSH (0.3-4.6 mU/L), 3) no history of structural heart disease, arrhythmia, or cardiac symptoms, 4) no history of comorbid diseases which affect thyroxine metabolism and cardiac structure, including hepatic or renal disease, anemia, and hypertension.Heart rate were evaluated at 2010 in control group.
comparison of N-terminal pro-brain natriuretic peptide (NT-pro-BNP) between groups | measure NT-pro-BNP at 2009 in DTC group and at 2010 in control group
  In DTC group, the investiagtors measured NT-Pro-BNP at 2009 (receiving TSH suppressive therapy for 5 to 9 years after thyroidectomy). As each DTC patient was enrolled, control subjects were selected from persons who visited endocrinology department for thyroid nodule work-up. The control group had to meet the following criteria: 1) the subject matched to a patient by age (±2 years), sex, and body mass index (BMI) (±2 kg/m2), 2) within the reference range of serum TSH (0.3-4.6 mU/L), 3) no history of structural heart disease, arrhythmia, or cardiac symptoms, 4) no history of comorbid diseases which affect thyroxine metabolism and cardiac structure, including hepatic or renal disease, anemia, and hypertension.NT-Pro-BNP was evaluated at 2010 in control group.
thyroid function test (TSH, free T4, free T3) | comparison of thyroid function at 2009 in case (DTC) and 2010 in control group
  In DTC group, the investiagtors measured thyroid function test at 2009 (receiving TSH suppressive therapy for 5 to 9 years after thyroidectomy). As each DTC patient was enrolled, control subjects were selected from persons who visited endocrinology department for thyroid nodule work-up. The control group had to meet the following criteria: 1) the subject matched to a patient by age (±2 years), sex, and body mass index (BMI) (±2 kg/m2), 2) within the reference range of serum TSH (0.3-4.6 mU/L), 3) no history of structural heart disease, arrhythmia, or cardiac symptoms, 4) no history of comorbid diseases which affect thyroxine metabolism and cardiac structure, including hepatic or renal disease, anemia, and hypertension.Thyroid function test was evaluated at 2010 in control group.

IPD SHARING:
Plan to Share IPD: No
We have no plan to share the data with other investigator.

REFERENCES:
- [Derived] Hong KS, Son JW, Ryu OH, Choi MG, Hong JY, Lee SJ. Cardiac Effects of Thyrotropin Oversuppression with Levothyroxine in Young Women with Differentiated Thyroid Cancer. Int J Endocrinol. 2016;2016:9846790. doi: 10.1155/2016/9846790. Epub 2016 Jun 23. PMID 27418929